CLINICAL TRIAL: NCT05226637
Title: Does Extra-corporeal Shock Wave Therapy Combined With Botulinum Toxin Type A Treatment Improve Clinical and Patient Reported Outcomes When Compared to Standard Management (BoNTA) in Patients With Upper Limb Spasticity of Cerebral Origin?
Brief Title: Does ESWT With BoNTA Treatment Improve Outcomes When Compared to Standard Management for Upper Limb Spasticity Patient.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00114513
Record Dates: First submitted 2021-12-23; First posted 2022-02-07 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Spasticity, Muscle
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: This two-arm parallel randomized double blinded controlled trial design study is designed as a pilot study, with the intention of using the result to inform a larger study across multiple centers. The study will be interventional using an existing device for specialized indication.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): In addition to standard of care, with BoNTA injections, the randomly selected control group will be treated with a sham head to the flexor muscles of the upper extremity. The sham component made by the manufacturers is designed such that the internal pneumatic projectile is physically blocked from providing high energy impact with the contact surface, however the handset looks and sounds identical. In doing so, the sham head still actuates and makes the same sounds but produces no shockwave
  ESWT will be apply on every candidate over the anterior region of the upper extremity injected with the BoNTA.
  Interventions: Device: Sham : The ESWT device (Storz Medical Duolith SD1),
- Experimental group with ESWT (Experimental): The randomly selected Study group will be comprised of patients who will receive the appropriate treatment with BoNTA in addition to actual ESWT (extra-corporeal shock wave therapy.
  ESWT is an existing technology that uses a device that generates high intensity shockwaves. These shock waves are generated outside of the body (extra corporeal) but penetrate through the skin surface to underlying structures and tissue. ESWT has been historically used safely and for many years to treat common musculoskeletal (MSK) conditions.
  For the purpose of the study these variables are standardized. We will treated with the Storz Duolith SD1 and we will use the D15 head 3000 number of shocks, 2.5 bar, 15 Hz over the same area of upper extremity described for the control group.
  Interventions: Device: ESWT (extra-corporeal shock wave therapy)

INTERVENTIONS:
Device: ESWT (extra-corporeal shock wave therapy) — The ESWT device (Storz Medical Duolith SD1),
  Arms: Experimental group with ESWT
Device: Sham : The ESWT device (Storz Medical Duolith SD1), — In doing so, the sham head still actuates and makes the same sounds but produces no shockwave. Because the patients receiving this intervention are naïve to ESWT, they will not be biased by the sensation it produces. Communication during treatment will be limited to avoid inadvertent bias.
  Arms: Control group

SUMMARY:
Background Effective management of spasticity, a debilitating and challenging condition afflicting many recovering from and living with neurological conditions, may reduce long term consequences such as limb contracture, skin breakdown, compromised mobility, caregiver burden and discomfort. In rehabilitation, spasticity represents a significant barrier to successful rehabilitation outcomes. Effective spasticity management can increases the length of individual functional status, reduces equipment/care needs, hospital admissions and extends the time people can stay safely at home, which would represent an economic benefit to the health system. Extra-corporeal Shock Wave Therapy (ESWT), an intense short energy wave delivered directly at the region of affected muscles has, in past randomized controlled studies, demonstrated positive outcomes for this population (spastic stroke population, TBI), on its own and as an adjunct to current modalities. In fact, one retrospective observational study demonstrated an increased efficacy of Toxin botulinum at 1 month when combined with ESWT. Where existing treatment options may be limited by coverage, access to delivery, complications and side effects, ESWT represents a potential to be a safe, low cost, efficacious alternative that can be administered by any trained clinician.

Aims The aims of this pilot study will be to explore the hypothesis that adding ESWT to Botulinum Neurotoxin A (BoNTA) in spasticity post-stroke (TBI)will demonstrate greater clinical and patient reported outcomes compared to standard treatment with BoNTA alone, a comparison only once previously studied.

Methods Incorporating randomization and placebo control (n= 20 in each arm), this patient-centric study will examine treatment goals and holistic perception of benefit after the treatment experience. We will use patient reported outcomes at baseline and at defined intervals after intervention. We will test our hypothesis using clinical and patient reported scales, such as the patient reported numeric rating scale (NRS) and goniometric range for spasticity as our primary outcome in conjunction with measures of muscle stiffness, quality of life, feasibility and acceptability of the protocol to help inform future study direction.

DETAILED DESCRIPTION:
Study Setting

The study will be performed within the Adult Spasticity Clinic at the Glenrose Rehabilitation Hospital (GRH) in Edmonton city in Canada. This is a dedicated space, appropriately equipped to support the safe treatment of spastic patients. Candidates will be recruited from our patient population and they will attend all appointments at the Spasticity Clinic. As a pilot project, we will be the only center involved in this study. The patient recruitment phase outlined in section 3.3 will identify agreeable participants. After successful enrollment there will be a series of 10-11 visits for the purpose of treatment, assessment and data collection. These visits are described in detail in appendix 1. The patient information and data will be collected by GRH Spasticity Program for Adults clinicians and stored in a secure location in accordance with the Health Information Act (Province of Alberta, 2000) and Freedom of Information and Protection of Privacy act (Province of Alberta, 2000).

Sample Size Determination

To adequately power this study a total of 20 participants for each group was calculated using the methodology advocated by Jones et al. (2003), An introduction to power and sample size estimation. This detail N value was calculated as follows:

Standardised difference = Difference between the means (Clinically important difference)/ Population standard deviation.

The clinically important difference as determined in a study by Farrar et al. (2008) is 1.27 for the Numeric Rating Scale for Spasticity. This is the difference that would detect a significant change in patient outcome. The standard deviation used was 2.0. This value was also to calculate the N value in their study. Therefore, according to this the standardized difference would be 1.27/2.0 = 0.635. When this is placed into Table 3 from Jones et al (2003) the number of patients needed to power this study would be approx. 54.4 pts (for a power level of 0.90) for a one-tailed hypothesis. As this study is a two-tailed hypothesis there would need to be double the patient numbers (54.4 X 2 = 108.8). Therefore, there would need to be approximately 109 patients enrolled in the study to adequately power it. Reflecting on the program's number of suitable patients with appropriate diagnoses and projected recruitment potential for the study, it was determined that a study of such magnitude could not easily be undertaken by a single site. For this reason, we have chosen to run this study as a pilot project. Based on these considerations a study population of 40 patients - 20 in each group was agreed to be an achievable target for our site. This pilot project would then help inform a larger study involving multiple centers.

Planning recruitment rate

The program holds treatment clinics for two full days per week with two physicians per day. The weekly patient numbers would total to between 30-40 appointments. Of these approximately 30% (9-12 patients) will typically be treated for spasticity of stroke origin. Another 10% (3 patients) will be patients with acquired brain injury from other sequelae, mainly traumatic brain injury and cerebral palsy. Given that the majority of these patients will have upper extremity spasticity with a MAS of 2 or more at the target joint, we may have a recruitment potential group of around 12-15 individuals per week. A conservative estimate will be that 75% of this number will have capacity to give consent, based on those who already consent for focal treatment, 9 to 11 individuals may have the potential to be enrolled. If the number of screened participants per week is 2, the recruitment rate would be 20 weeks. An additional 10 weeks could reasonably add to accommodate for recruitment variances, screen failure and drop out top achieve the sample size of 40 participants.

Recruitment strategy

As the only program providing complex spasticity management in the locale in sufficient numbers, the participant population will be recruited directly from the Spasticity Program for Adults program at the GRH, no external advertising will be required. The seven program physicians, understanding the inclusion/exclusion criteria will provide pre-screen selection for potential participants. Interested individuals will then be provided with an information sheet including contact numbers for the research team. Interested patients may then call the Program RN (study coordinators) for more information or to enroll for initial screening and, if appropriate, informed written consent will then be obtained to participate in the study. (See written consent sheet annexe 2. It will be also stressed that at any time, the participant can exercise his or her right to withdraw from the study without prejudice and be free to continue his or her pre-existing spasticity management.

It is estimated that he likely rates of loss to follow up is low considering all participants will continue to receive standard care within the clinic and would be motivated to receive treatment that may provide a greater degree of relief from spasticity. Treatment discomfort, however, may contribute to attrition if it is found to be more noxious than anticipated or adverse events have caused participants to withdraw. For this reason, we would reserve the right to enroll a further 10 candidates to achieve the target of 40 participants completing the study.

Recruitment time period

The recruitment time period should be over a period of 4-6 months. Taking into consideration that most of our injection patients are seen on a four months cycle. This will allow us to capture a large majority of our existing patients through their injection's cycles.

Criteria for Discontinuing or Modifying Interventions

Treatment will be withdrawn at any time at the participant's request. If the participant feels that shockwave treatment is not suitable or has demonstrated an adverse reaction to which they feel uncomfortable to proceed, they will be removed from the study at their request. Any of the clinicians on the team can also remove the patient from the study at any time if it is demonstrated that they are having a detrimental adverse reaction to the treatment. All adverse events and causes will be documented and with any actions taken as well as final disposition. Adverse events deemed to be serious (unforeseen injury) will be reported immediately to the responsible physician and any follow up documented. Missed appointments will be documented and if possible, the cause identified. Failure to adhere to the appointment schedule will result in withdrawal from the study. Given the complexity of appointment planning an appointment schedule modification of +/- one day will be allowed in extenuating circumstances and will be subject to the research group's availability.

Concomitant care and interventions

Participants are allowed to maintain their current level of therapy but will not be permitted to add any new interventions during the study period. Participants are allowed to maintain their current medications but will not be permitted to change any anti-spasticity medication that may affect assessments. If the responsible physician deems medication changes as necessary, then that participant will be removed from the study.

The sources of data will be:

Historical: Participant Screening Form identifying:

* Participant number
* It will allow us to anonymously identify the participant in throughout the study.
* Sex
* For purpose of stratification and analyze.
* Age or year of birth
* For purpose of stratification and analyze.
* Primary Diagnosis
* It is necessary for inclusion criteria since the spasticity must be secondary to brain lesion.
* Area/s affected by spasticity
* Must necessarily have elbow flexor increase tone. It is also mandatory to know which muscles to treat.
* Medical History
* To avoid complication or counterindication of the treatment.
* Current Medication
* We need to know any medication used for spasticity, pain or mood disorder since it can influence the response to the focal treatment dispensed and influence answers on different questionnaires and scales. We also need to know if they are taking medication to lighten the blood which can increase to risk of bleeding post injection or ESWT.
* Applicable INR History
* I it is too high; it will increase the risk of bleeding post injection or ESWT.
* Contraceptive method
* It is part of our inclusion/exclusion criteria.

Patient Reported Outcomes:

* NRS spasticity,
* NRS pain,
* EQ-5D-5L

Clinical outcomes:

* Physical assessment of target limb MAS,
* Passive ROM of elbow,
* Which muscles injected with BoNTA and the numbers of muscles injected, with which toxin and the number of units used
* Applicable pregnancy test if needed
* INR tests if needed

Statistical Methods.

Demographic, comorbidities and other contextual data will be collected, and descriptive statistics will be used to summarize these data along with other variables including passive range of motion (PROM) at the affected elbow and MAS and responses to patient reported outcome data (PRO) such as the EQ5D-5L. Median and inter-quartile ranges will be reported for all data due to the likely skewed distribution resulting from the small sample size.

Pre and post intervention paired data on NRS, PROs will be compared using the Wilcoxon signed-rank test. For the PRO data two-tailed test will be used and a p<0.05 considered significant. For the NRS, the clinically important difference for improvement in the NRS has been reported to be a mean difference of 1.27 with a SD of 2.0 (Farrar et al. 2008 and Collin et al 2010) two tailed test will be used to detect any improvement or deterioration in spasticity.

Correlations will be examined between MAS, NRS and PROM scores using Spearman Rank correlation coefficients. For the EQ5D-5L descriptive data will be reported for the five component dimensions and VAS summary overall health. The index utility score for the EQ5D-5L health states will be calculated based on the Canadian population-based preference weights (Xie et al 2016). Differences between the groups will be analyzed using the Mann-Whitney test. Multiple logistic regression will be used to predict improvement in spasticity based on demographic and other contextual data. In order to check for association between the variables entered into the model the correlation matrix will be examined for high values of pair-wise correlations and a value of >0.8 considered to indicate potential multicollinearity (Grewal et al 2004)

ELIGIBILITY:
Inclusion Criteria:

* People with upper limb Spasticity of Cerebral Origin, including but not limited to:
* Acquired brain injury (of at least 1 year following the event);
* Stroke;
* Cerebral Palsy (CP);
* Male and females over 18 years of age.
* Female subjects must either be post-menopausal, sterilized (at least 12 months post menses) or be consistently using a highly effective method of birth control such as a sterilized partner, oral/implanted/injected contraception or abstinence of sexual activity and be willing to provide a pregnancy test as the safe use of ESWT during pregnancy has not been demonstrated.
* Being naive to shockwave therapy;
* Spasticity as defined by Modified Ashworth Scale (MAS) score of 2 in a functional or non-functional upper limb affecting the target joint, which for the purpose of the study will be the elbow;
* Willingness to participate and provide written consent;
* Have the cognitive capacity to answers simple questionnaires;
* Either already receiving treatment with BoNTA and having been 'washed out' for a period of three months, or intends to begin 'standard treatment with BoNTA to an affected arm with target joint involvement.
* Standard treatment in the context of the study will include, in addition to any other therapies, focal treatment with Botulinum Neurotoxin Type A to treat the target joint.

Exclusion Criteria:

* Known neurodegenerative disorder at the spinal level;
* Known spinal cord lesion ;
* Fixed contracture of target joint impeding assessment or MAS of 4;
* Any demonstrated lower motor neuron damage to the affected limb;
* Surgery received to affected arm that may affect assessment of the target joint;
* Any changes in either oral or focally injected medications one month prior to screening to close out, that could influence any outcome measures;
* Any changes in medication one month prior to screening to close out, for the treatment of depression as changes in patient affect may influence outcome measures;
* Any changes in rehabilitation therapy throughout the study cycles;
* Confirmed pregnancy. Safe use in this population remains unknown;
* Nursing mothers. Safe use in this population remains unknown;
* Female patients who are of childbearing age without adequate contraception and unwilling to take a pregnancy test;
* Implanted electronic device/s. Kinetic energy in the same territory as an implanted device may adversely affect the device's function;
* Patients taking Warfarin and have poorly controlled coagulopathy or an INR above 3 at the Point of Care. To avoid hematoma, compartment syndrome or other consequences of prolonged bleeding to treated area. This is also the same program criteria for injection with BoNTA. For this population INR will be determined (using the Coguchek XL device) prior to each treatment;
* Any malignant diagnoses. Tissue disruption caused by the shockwave treatment may precipitate the liberation or shedding of cancer cells;
* Any known infection, inflammatory process, open areas or acute undiagnosed swelling (acute being defined as 14 days or sooner) in the area treated to avoid worsening of any pre-existing condition;
* Participation in any other concurrent study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in patient reported outcomes of spasticity on Numerical Rating Scale (NRS) for Spasticity at weeks 4, 12 and 24. | 4, 12 and 24 weeks from the baseline
  The primary patient reported outcome will be the Numerical Rating Scale (NRS) for Spasticity This is a 0-10 scale where the patients rate their spasticity over a 24hr period. Spasticity in this context is defined to the patients as the experience of muscle stiffness at the target joint over this specified period of time. (farrar et al). The NRS when used in spasticity has been shown to be valid and reliable by farrar et al 2008. It was also shown to correlate with objective scores such as the Modified Ashworth and Tardieu Scales for directly assessing spasticity at a given joint. This study also confirmed that the NRS for Spasticity is a reliable and valid tool in the assessment of spasticity. (Anwar and Barnes, 2009).
Change from baseline in clinical passive range of motion at the elbow joint treated side with goniometer at weeks 4, 12 and 24. | 4, 12 and 24 weeks from the baseline
  The primary clinical outcome will be the passive range of motion available at the elbow on treated side with a goniometer. It is an instrument that either measures an angle or allows an object to be rotated to a precise angular position. These measurements help accurately track progress in a rehabilitation program. At the elbow, the axis location will be on lateral epicondyle, the stationary arm parallel with the humerus and the movement arm of the goniometer parallel with the radius. Usually, the normal Range of motion at the elbow is around 150 degrees

SECONDARY OUTCOMES:
Change from baseline of patient reported outcomes quality of life on EQ-5D-5L questionnaire at weeks 4, 12 and 24. | 4, 12 and 24 weeks from the baseline
  The secondary patient reported outcome will be the EQ-5D-5L. It is a validated five dimensional quality of life questionnaire recording variance using a five points scale to determine the participant's self-perception of mobility, self-care, usual activities, pain/discomfort, anxiety/depression
Change from baseline on spasticity level on Modified Ashworth Scale (MAS) at 4, 12 and 24 weeks | 4, 12 and 24 weeks from baseline
  The secondary clinical outcomes variables will be the Modified Ashworth Scale (MAS) provides a simple, validated and easily replicable method of assessing objectively the participants level of spasticity in the target joint. This will be compared with the NRS to support correlation between the subjective and objective nature of the two assessment tools.

OTHER OUTCOMES:
Feasibility of the project measured by the percentage of participants without any missing data at the end of the study and percentage of participant who completed the study. | 24 weeks
  Feasibility of the project will be mainly determine by the adherence to the protocol. To measure it we will use:
  1. Percentage of number of participants without any missing data at the end of the study (all measurements and questionnaires have be done and recorded).
  2. Percentage of number of participants who drop-out of the study at the end of the study.
Measure the acceptability of the procedure (ESWT) throughout the study using a pain numerical rating scale (NRS). | once a week for 3 weeks at ESWT therapy
  Acceptability of the procedure, defined as the extent to which participants considered ESWT reasonable and appropriate in terms of their experience.
  We will use : measured as self-reported symptoms of pain during each of the assessments using a numerical rating scale ranging from 0 [no discomfort] to 10 [worst pain imaginable]

CONTACTS AND LOCATIONS:
Overall Officials: Lalith E Satkunam, MD, Principal Investigator — Alberta University
Locations (1):
- Glenrose Rehabilitation Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
no plan